CLINICAL TRIAL: NCT02649530
Title: An Open Label, Non-randomized Phase II Trial Evaluating WNT974 in Patients With Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Phase II Trial Evaluating WNT974 in Patients With Metastatic Head and Neck Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding withdrawn
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.157; HUM00108169 (Other: University of Michigan)
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Squamous Cell Carcinoma, Head And Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — LGK974

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WNT974 (Experimental): Patients will receive 10 mg of WNT974 daily by mouth.
  Interventions: Drug: WNT974

INTERVENTIONS:
Drug: WNT974

SUMMARY:
Given that up-regulation of the Wnt pathway has been identified as having a significant role in carcinogenesis in advanced head and neck squamous cell carcinoma, the investigator believes that inhibition of Porcupine via WNT974 will result in tumor control hence improvement in disease free and overall survival in these patients with a tolerable toxicity profile. As suggested by pre-clinical models, patients with a tumor harboring a Notch receptor (any of the four) loss of function mutation may have a greater response rate to treatment with WNT974. The investigator aims to address this question by administration of single agent WNT974 and following response radiologically along with close clinical follow up to monitor toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of locally advanced or metastatic SCC (Squamous Cell Carcinoma) of the head and neck no longer amenable to curative surgical resection or radiation therapy.
* Refractory to platinum-based therapy (defined as disease progression within 6 months of last dose of platinum chemotherapy)
* Patient is able swallow and absorb oral medications
* Age 18 years or older
* ECOG Performance Status (an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death) of 0-2
* Patients must have CT (CAT Scan) measurable disease as defined by RECIST v1.1
* Willingness and ability to comply with all study procedures
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.
* Archival tissue available for Foundation One analysis.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.

Exclusion Criteria:

* Inability to obtain Foundation One testing on archival tissue, or, lack of previous Next Generation Sequencing incorporating testing for NOTCH -1, -2, -3, and -4
* Impaired cardiac function including any one of the following:
* Patients with any of the following laboratory values at baseline: Absolute neutrophil count (ANC) < 1,000/mm3 [SI units 109/L], Platelets < 75,000/mm3 [SI units 109/L], Hemoglobin < 9.0 gm/dL [SI units gm/L], Calculated (e.g. using Cockcroft-Gault formula) or measured creatinine clearance < 50 ml/min, Bilirubin > 1.5 x ULN, except for patients with known Gilbert syndrome who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN, Aspartate transaminase (AST) > 3.0 x ULN, except for patients with liver metastasis who are excluded if AST > 5.0 x ULN, Alanine transaminase (ALT) > 3.0 x ULN, except for patients with liver metastasis who are excluded if ALT > 5.0 x ULN
* Impairment of GI function or GI disease that may significantly alter the absorption of WNT974
* Presence of ≥ CTCAE (Common Terminology Criteria for Adverse Events) Grade 2 toxicity (except alopecia) due to prior therapy
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion criterion include the following: malignancies that were treated curatively, and have not recurred within 3 years prior to study entry; completely resected basal cell and squamous cell skin cancers; and completely resected carcinoma in situ of any type
* Patients who received anti-cancer therapy prior to the first dose of WNT974 within the following time frames: Biological therapy with a prolonged half-life (e.g., monoclonal antibodies) within 4 weeks, Cytotoxic agents associated with delayed hematologic recovery (e.g., nitrosourea or mitomycin-C) within 6 weeks, Other systemic anti-cancer agents within 3 weeks, Radiotherapy within 2 weeks
* Patients who are currently receiving treatment with medications that meet one of the following criteria and that cannot be discontinued at least one week prior to the start of treatment with WNT974: Strong inhibitors or inducers of CYP3A4/5, CYP3A4/5 substrates with narrow therapeutic index, known to prolong the QT interval and are also CYP3A4/5 substrates. Refer to Appendix 1 for guidance on concomitant medication.
* Patients who have undergone any major surgery within 2 weeks prior to starting study drug or who have not adequately recovered from previous surgery
* Active hepatitis B or C infection
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 30 days after study treatment. Highly effective contraception methods include: Total abstinence or, male or female sterilization, combination of any two of the following: Use of oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception. Post-menopausal women are allowed to participate in this study.
* Sexually active males must use a condom during intercourse while taking the drug and for 90 days after stopping treatment and should not father a child in this period.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation
* Patients residing in prison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The number of patients with stable disease, complete response and partial response | 4 months
  Disease control rate will be assessed by examining the number of patients with stable disease, complete and partial response.

SECONDARY OUTCOMES:
Number of patients that respond to treatment | 4 months
  The overall response rate will be determined. Overall response will be defined as the sum of complete response + partial response.
Duration of time from start of treatment to time of progression | 6 months post treatment
  Progression free survival in patients with metastatic head and neck cancer will be determined.
The number of patients alive at 6 months post treatment | 6 months post treatment
  Overall survival will be examined.
The number of patients that experience adverse events | 4 weeks post treatment
  Toxicities associated with the treatment of WNT974 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Worden, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States